CLINICAL TRIAL: NCT05323253
Title: A Prospective International Multicenter, Pivotal, Single Arm, Open Label Clinical Study to Assess the Efficacy and Safety of Intratumoral Alpha DaRT224 for the Treatment of Patients With Recurrent Cutaneous Squamous Cell Carcinoma
Brief Title: A Clinical Study to Assess the Efficacy and Safety of Alpha DaRT224 for the Treatment of Patients With Recurrent Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-SCC-03
Record Dates: First submitted 2022-04-01; First posted 2022-04-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma; Recurrent Squamous Cell Carcinoma; Alpha emitting radiation; Carcinoma, Squamous; Skin Cancer; Brachytherapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an International Multicenter, Pivotal, Single Arm, Open Label pivotal trial with DaRT for the treatment of Recurrent Cutaneous Squamous Cell Carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- DaRT seeds (Experimental): DaRT source will be inserted using preplanned radiotherapy parameters and reassessed by volumetric imaging 2-3 weeks after placement and then removed. Objective Response Rate (ORR) will be determined based on confirmed BOR following DaRT insertion.
  Interventions: Device: DaRT seeds

INTERVENTIONS:
Device: DaRT seeds — DaRT source will be inserted using preplanned radiotherapy parameters and reassessed by volumetric imaging 2-3 weeks after placement and then removed.
  Other Names: DaRT

SUMMARY:
This is a multi-center clinical study enrolling up to 86 participants. The primary objectives are to determine the objective response rate (ORR) established by the confirmed best overall response (BOR) following intratumoral administration of DaRT - Diffusing Alpha-Emitters Radiation Therapy, as well as to assess the Duration of Response (DOR) 6 months from initial response. Secondary objectives are to assess the safety of DaRT, and to assess the progression free survival (PFS), overall survival (OS), Overall Duration of Response (O-DOR), local control and quality of life (QOL) for patients treated with DaRT.

DETAILED DESCRIPTION:
This study is a prospective multicenter, pivotal, single arm, open label clinical study to assess the efficacy and safety of intratumoral Alpha DaRT-224 for the treatment of patients with recurrent cutaneous squamous cell carcinoma.

The "Diffusing Alpha-emitter Radiation Therapy (DaRT)", based on the interstitial intratumoral placement of an encapsulated Radium-224 source (3.7 days half-life), is described in this study. These sources release short-lived alpha-emitting atoms into the tumor microenvironment by recoil. DaRT seeds will be inserted into recurrent Squamous Cell Carcinoma (SCC) tumors and will be removed following 14-21 days.

The Objective Response Rate (ORR) will be determined based on the confirmed Best Overall Response (BOR) following DaRT insertion. Duration of Response (DOR) will be assessed for up to 6 months from initial response is documented. Safety will be assessed based on the cumulative incidence rate, severity and outcome of device related Adverse Events (AEs). Classification of AEs will be done according to CTCAE v5.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent cutaneous SCC histologically confirmed who have failed at least first line standard of care therapy who are not indicated for surgery and standard radiation therapy, or non alpha radiation brachytherapy technologies, and for whom no curative systemic treatment is available
2. Central histopathological confirmation within 6 months of enrollment provided no tumor treatment occurred between the biopsy and enrollment
3. Measurable disease according to RECIST v 1.1.
4. Ability to undergo a CT scan
5. Tumor size ≤7 cm, at the longest diameter.
6. Single lesion per subject.
7. Targeted lesion must be technically amenable for complete coverage (including margins) by the DaRT seeds.Targets will be deemed technically amenable for complete coverage if there are entry and exit vectors for placement that are not hindered by bone or major vessels or other vital organs (eg. eye).
8. Interstitial implant indication validated by multidisciplinary team.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
10. Life expectancy ≥12 months.
11. Subjects male/ female ≥18.
12. Willing and have the ability to provide signed Informed Consent.
13. Patients, male and female, with reproductive potential (including women who are menopausal for less than a year and not surgically sterilized), must practice acceptable effective methods of birth control, such as barrier methods, condom or diaphragm with spermicide or abstinence. Birth control should be continued for 3 months after the DaRT insertion visit.
14. Women with childbearing potential must provide a negative pregnancy test during the screening period and up to V1, prior to the DaRT insertion procedure.
15. Blood tests values:

    * Leucocytes ≥3000mm3,
    * Absolute neutrophil count ≥1500mm3,
    * Platelets ≥100,000 mm3,
    * Total bilirubin ≤ 1.5xULN (upper limit of normal)
    * Aspartate Aminotransferase (AST) ≤2.5xULN,
    * Serum Glutamic-Oxaloacetic Transaminase (SGOT) ≤2.5xULN,
    * Serum Glutamic-Pyruvic Transaminase (SGPT) ≤2.5xULN,
    * Alkaline Phosphatase ≤2.5xULN.
    * Creatinine ≤ 2.0xULN or Creatinine Clearance ≥60 ml/min.
    * INR (International Normalized Ratio) or Prothrombin time ≤1.5xULN.

Exclusion Criteria:

1. Distant or nodal metastatic disease (according to the TNM [tumor, nodes , and metastases] staging system - N+ or M1 patients are excluded).
2. T4 disease or perineural spread of disease
3. Previously untreated cutaneous SCC indicated for surgery or radiation.
4. Mucosal, vulvar, anal and penile SCC.
5. Inability to fully cover the entire volume with DaRT seeds
6. Inability to place DaRT seeds into tumor due to inaccessibility by presence of bones or major vessels or vital organs
7. Inability to undergo a CT scan
8. Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
9. Patients receiving any of the following within 4 weeks of enrollment:

   1. Antineoplastic systemic chemotherapy or biological therapy
   2. Immunotherapy
   3. Investigational agents other than the study intervention
   4. Radiation therapy
   5. Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial.
10. Longest tumor diameter >7 cm.
11. Tumor with keratoacanthoma histology.
12. Known hypersensitivity to any component of treatment.
13. Clinically significant cardiovascular disease e.g., cardiac failure of New York Heart Association class III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, history of myocardial infarction in the last 12 months.
14. Any medical or Psychiatric illness, which in the opinion of the investigator would compromise the patient's ability to tolerate treatment and to adhere to the clinical trial protocol.
15. Serious medical comorbidities that, in the opinion of the investigator, may affect subject compliance and/or interpretation of treatment safety or effectiveness.
16. High probability of protocol non-compliance (in opinion of investigator).
17. Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
18. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
19. Patients do not agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry and for 3 months after the DaRT insertion visit.
20. Breastfeeding or pregnant women
21. Tattoos or other identifying marks which can not be adequately hidden on digital photos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From Day 14 until 52 weeks
  Objective Response Rate (ORR) of DaRT as treatment for Recurrent SCC established by the confirmed Best Overall Response (BOR), with confirmation at least 4 weeks after initial assessment
Duration of Response | 6 months from from first demonstration of CR or PR after Alpha DaRT seeds insertion.
  Assess the Duration of Response (DOR) of DaRT as treatment for Recurrent SCC

SECONDARY OUTCOMES:
Progression Free Survival | Up to 12 months after DaRT seed insertion
  Determine Progression Free Survival (PFS) of SCC following DaRT treatment
Overall Survival | Up to 12 months following DaRT insertion
  Assess Overall Survival (OS) of Recurrent SCC patients treated with DaRT
Time of Local Control | Up to 12 months following DaRT insertion
  Local control of SCC following DaRT treatment is measured as the time from first recorded response (Complete Response/Partial Response/Stable Disease) to local recurrence up to 12 months or last follow up
Patients Quality of Life Assessment | On 14 days,12 weeks and 52 weeks following DaRT insertion
  Assess patient reported health related quality of life (QOL) outcomes using the Skin Cancer Index (SCI) and Skindex-16 questionnaires
DaRT-related Adverse Events | Up to 12 months following DaRT insertion
  Assess the safety of the Alpha DaRT treatment, based on the cumulative incidence rate, severity and outcome of device related AEs. Classification of AEs will be done according to CTCAE v5
Overall Duration of Response (O-DOR) | Up to 12 months following first reported response
  O-DOR Defined as the time from first response (CR or PR) to the date of initial objectively documented progression or death due to any cause, whichever occurs first.
User experience | On Day 0 (DaRT insertion) and Day 14 (+7) (DaRT removal)
  Assess user experience as determined by questionnaire

CONTACTS AND LOCATIONS:
Locations (30):
- United States (25):
  - Banner Health MD Anderson Phoenix, Gilbert, Arizona
  - Dignity Health Cancer Institute, Phoenix, Arizona
  - Alliance Dermatology, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - Day Star Skin and Cancer Center, DeLand, Florida
  - Integrity Research Clinical Associates, Delray Beach, Florida
  - Palm beach Dermatology Group, Delray Beach, Florida
  - Hollywood Dermatology, Hollywood, Florida
  - University of Miami, Miami, Florida
  - Baptist Health South Florida MCI, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Beer Dermatology, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Schweiger Dermatology Group, Hackensack, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Bassett Healthcare Network, Cooperstown, New York
  - Northwell Health, Queens, New York
  - New York Medical Skin Solutions, Rockaway Park, New York
  - MDCS Dermatology, Smithtown, New York
  - West Cancer Center, Germantown, Tennessee
  - Gulf Coast Cancer Center, Houston, Texas
  - University Cancer & Diagnostic Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Dermatology of Seattle and Bellevue, Bellevue, Washington
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Belinson-Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan